CLINICAL TRIAL: NCT04873414
Title: Clinical Trial of Convalescent Plasma Administration as Adjunct Therapy for COVID-19 (Uji Klinik Pemberian Plasma Konvalesen Sebagai Terapi Tambahan COVID-19)
Brief Title: Convalescent Plasma as Adjunct Therapy for COVID-19
Acronym: PlaSenTer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Health Research and Development, Ministry of Health Republic of Indonesia (Other)
Collaborators: Indonesian Red Cross (Unknown); Eijkman Institute for Molecular Biology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVID-CT002
Record Dates: First submitted 2021-04-26; First posted 2021-05-05 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: COVID-19
Keywords: COVID-19; Moderate; Severe; Convalescent Plasma; Indonesia
MeSH Terms: conditions — COVID-19; Lymphoma, Follicular | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Subjects in the Treatment Group are given 200 ml of Plasma collected from Convalescent Patients recovered from COVID-19 at two-day intervals in addition to standard supportive treatment
  Interventions: Biological: Convalescent plasma treatment
- Control group (No Intervention): Subjects in the Control Group are given standard supportive treatment

INTERVENTIONS:
Biological: Convalescent plasma treatment — Convalescent Plasma collected from patients who recover from COVID-19 and have been discharged from the hospital for at least 14 days.
  Arms: Treatment group

SUMMARY:
Convalescent plasma (CP) has been the subject of increasing expectation for treating coronavirus disease 2019 (COVID-19). Reports on CP transfusion have shown promising clinical improvements without serious adverse events. To date, most studies focused on reporting CP treatment in patients with severe COVID-19, but only a few addressed benefits on less severe disease. The vast majority of studies reporting COVID-19 infection and treatment have come from earlier affected countries with established health systems and research infrastructure, while very few are from low- and middle-income countries (LMICs). Nonetheless, CP therapy could be one of the few available options in LMICs where constraints may exist in the access to novel treatments, even once available. Clinical trials conducted in LMICs may differ in many respects from those in high-income countries.

This study will evaluate the safety and efficacy of convalescent plasma therapy in hospitalized with moderate and severe COVID-19, to investigate the impacts of the treatment over the course of clinical illness, including non-mortal clinical outcomes.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19), which is caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), has spread rapidly around the world, with high rates of transmission and substantial mortality.

Convalescent plasma (CP) collected from recovered patients has been evaluated in the treatment of SARS, Middle East respiratory syndrome (MERS), and Ebola, but not well further studied and with no definitive results. Preliminary studies in COVID-19 patients showed improvement in clinical status after CP transfusion. However, a multicenter, open-label, randomized clinical trial of 103 patients in China with severe or life-threatening COVID-19 found no statistical difference in clinical improvement within 28 days among patients treated with CP versus standard treatment alone.

To date, CP has not been approved as a standard of care for COVID-19. There are insufficient data from well-controlled, adequately powered, randomized clinical trials to evaluate the efficacy and safety of CP for the treatment of this disease. One randomized controlled trial (NCT04342182) was halted for redesign based on the consideration that most COVID-19 patients already have high neutralizing antibody titers at hospital admission and no difference in mortality (p=0.95), hospital stay (p=0.68), or day-15 disease severity (p=0.58) was observed between plasma treated patients and patients on standard of care. Another clinical study (NCT04345523) showed efficacy and safety of CP in preventing progression to severe disease or death. However, this study was halted early due to low enrolment. Further studies have been published and assessed in several systematic reviews that remain uncertain about the safety and effectiveness of CP treatment for COVID-19.

The vast majority of studies reporting COVID-19 trials have come from the earlier affected countries with established healthcare systems and better research infrastructure, while very few are from low- and middle-income countries (LMICs). Meanwhile, the cases in LMICs have risen considerably with critical research questions specific to the needs of are hard to answer. As an LMIC with a geographically dispersed archipelago, access to healthcare remains a challenge in remote districts that could impact the adoption of CP deployment in Indonesia. Consequently, clinical trials conducted in LMICs may differ in many respects from those in high-income countries.

This study will evaluate the safety and efficacy of CP therapy in hospitalized with moderate and severe COVID-19, to investigate the impacts of the treatment over the course of clinical illness, including non-mortal clinical outcomes. This study will involve hospitals from different places of the Indonesian archipelago, with different characteristics and community structures, social, and values. To obtain supports for the trial, the investigators will seek community engagement that allows investigators and community leaders working collaboratively.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Patients with PCR-confirmed COVID-19
2. Minimal age:18 years
3. Agree to participate in the trial with written informed consent
4. Moderate or Severe COVID-19 at the time of enrollment

   .

   A. Definition of moderate disease (according to Siddiqi et al):

   Moderate COVID-19 is defined as disease with fever, respiratory symptoms (dry cough, chest distress, or shortness of breath after activities), and pulmonary imaging findings, and at least one of the following findings:

   i) Abnormal coagulation parameters:
   * D-dimer >1 µg/mL (normal <0.5 µg/mL)
   * Prothrombin time (>13.6 second) or International normalized ratio (INR) ≥1.8
   * Thrombocyte count <100x 10^3/mL

   ii) Increased pro-inflammatory markers:
   * C-reactive protein (CRP) ≥26.9 mg/L
   * Procalcitonin ≥0.5 ng/mL,
   * Lymphocyte count <1.5x 10^9/L) or Neutrophil/Lymphocyte ratio (NLR) >3.3

   iii) Presence of risk factors or comorbidities:
   * Age >65 years
   * Type 1 Diabetes Mellitus or type 2 Diabetes Mellitus (with any of the following: Fasting blood glucose ≥126 mg/dl, 2-h plasma glucose ≥200 mg/dL, or random plasma glucose ≥200 mg/dL, plus HbA1C >6.5%)
   * Chronic kidney disease (creatinine >2.0 mg/dL) or with routine hemodialysis
   * Chronic liver Disease with signs of liver cirrhosis; Child-Turcotte-Pugh (CTP) Class A (score 5-6) or Class B (score 7-9) or higher; or Model for End-Stage Liver Disease (MELD) score <39
   * Heart failure (New York Health Association [NYHA] Class I or II)
   * Bronchial asthma, chronic obstructive pulmonary disease (COPD), or pulmonary tuberculosis
   * Cancer (particularly patients with chemotherapy or immunotherapy)
   * Immunocompromised conditions, including HIV/AIDS, post-organ transplantation, or judged by attending physician (preferable after specialist consultation)
   * Long-term corticosteroid use
   * autoimmune disease
   * Sequential Organ Failure Assessment [SOFA] score ≥5.65
   * Body Mass Index (BMI) ≥35 kg/m2

   B. Definition of severe COVID-19 (according to Siddiqi et al):

   Severe Covid-19 is defined as disease with a respiratory rate ≥30 breaths/min, oxygen saturation <90% or oxygenation index (PaO2/FiO2) ≤300 mmHg, and/or lung infiltrates >50% within 24-48 h.

   EXCLUSION CRITERIA:
   * Pregnant or lactating woman
   * History of transfusion reaction, blood-group incompatibility, IgA deficiency, or Allergy to Immunoglobulin-containing substances
   * Concurrent participation of clinical trials of COVID-19 treatment
   * Possibility of transfer to other hospital within 72 hours
   * Heart Failure (NYHA Class III or higher) or other diseases with risks of volume overload
   * Permanent organ failure unrelated to COVID-19, including:

     * End-stage liver disease (CTP score >10 or MELD score >40)
     * End stage renal disease with creatinine clearance <30% or in routine dialysis
   * Multiple organ failure (SOFA score ≥11)
   * Concomitant condition or treatment with risks of thrombosis, e.g., cryoglobulinemia, refractory hypertriglyceridemia, or monoclonal gammopathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 364 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The mortality in COVID-19 patients treated with convalescent plasma | From the initiation of CP treatment until hospital discharge or death, up to 28 days
  Number of deaths from the initiation of CP treatment until hospital discharge or death.

SECONDARY OUTCOMES:
Change in clinical status category in CP-receiving patients | From the initiation of CP treatment until hospital discharge or death, up to 28 days
  Change in clinical status category will be scored daily based on the modified WHO six-point ordinal scale. The six-point scale is as follows: 1, non-hospitalized; 2, hospitalized, without supplemental oxygen; 3, hospitalized, with supplemental oxygen; 4, hospitalized, with nasal high-flow oxygen therapy, non-invasive mechanical ventilation, or both; 5, hospitalized, with invasive mechanical ventilation, extracorporeal membrane oxygenation (ECMO), or both; and 6, death
Duration of hospitalization | From admisstion until hospital discharge or death, up to 28 days
  Number of days from the admission to the date of discharge or death. Patients who are not discharged and remain in the hospital at the end of study period will be censored on the study's end date, while those who are lost to follow-up will be censored on the last encounter date
Duration of mechanical ventilation | From the initiation of CP treatment until hospital discharge or death, up to 28 days
  Number of days in patients with ventilatory support
Duration of ICU stay | From the initiation of CP treatment until hospital discharge or death, up to 28 days
  Number of days from entry to release from ICU
Change in lung image radiography in CP-receiving patients | Days 0, 6, 14, 21, and 28
  The lung radiological image will be assessed using the Brixia chest X-ray scoring (Morghesi and Maroldi, 2020). Each lung is divided into three zones, marked by letters A, B, and C for the right lung, and D, E, and F for the left lung. The letters divide the lungs into three levels: upper level (A and D), above the inferior wall of the aortic arch; middle level (B and E), below the inferior wall of the aortic arch and above the inferior wall of the right inferior pulmonary vein; and lower level (C and F), below the inferior wall of the right inferior pulmonary vein. A score (from 0 to 3) is assigned to each zone based on the detected lung abnormalities: 0, no lung abnormalities; 1, interstitial infiltrates; 2, interstitial and alveolar infiltrates (interstitial pre-dominance); and 3, interstitial and alveolar infiltrates (alveolar predominance). The overall CXR score is the sum of points from the six lung zones with a range from 0 to 18.
Change in inflammatory parameters in CP-receiving patients | Days 0, 6, 14, 21, and 28
  Measurement of C-reactive protein (reference: <5.0 mg/L); neutrophil/lymphocyte ratio reference range: male, 0.43~2.75; female,0.37~2.87), procalcitonin (reference: <0.15 ng/mL), and IL-6 (reference range: (5-15 pg/ml) levels in CP-receiving patients
Change in coagulation parameters in CP-receiving patients | Days 0, 6, 14, 21, and 28
  Measurement of D-Dimer (reference: <0.5 mcg/mL) and prothrombin time (reference range: 11.0-13.6) seconds in CP-receiving patients
Change in viral load in CP-receiving patients | Days 0, 3, 6, 14, 21, and 28
  Measurement of viral load by nasopharyngeal swab PCR in CP-receiving patients. Additional test on day 3 will be performed to identify the early clearance of the virus.
Changes in anti-SARS-CoV-2 antibody levels in CP-receiving patients | Days 0, 3, 6, 14, 21, and 28
  Plasma/serum titer of anti-SARS-CoV-2 antibodies in CP-receiving patients by the plaque reduction neutralization test or enzyme-linked immunosorbent assay. Additional test on day 3 will be performed to identify the early changes in antibody levels.
Systemic organ involvement in patients receiving CP treatment | Days 0, 6, 14, 21, and 28
  Systemic organ involvement measured by the Sequential Organ Failure Assessment (SOFA) score. It is used for calculation of both the number and the severity of organ dysfunction in six organ systems (respiratory, coagulatory, liver, cardiovascular, renal, and neurologic), and can measure individual or aggregate organ dysfunction. Each organ system is assigned a point value from 0 (normal) to 4 (high degree of dysfunction/failure). The SOFA score ranges from 0 to 24. An increasing or unchanged SOFA score is associated with a higher mortality rate than patients with a decreasing score.
Time to resolution of symptoms in patients receiving CP treatment | Days 0, 6, 14, 21, and 28
  Patients whose symptoms are not resolved and remain in the hospital at the end of study period will be censored on the study's end date, while those are lost to follow-up will be censored on the last encounter date.
Treatment-related adverse events (AEs) and serious adverse events (SAEs) | From the initiation of CP treatment until hospital discharge or death, up to 28 days
  Number of participants with treatment-related adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Impact of anti-SARS-CoV-2 antibody levels in donors on the efficacy of CP therapy in CP-receiving patients | Days 0, 6, 14, 21, and 28
  Correlation between anti-SARS-CoV-2 antibody levels in donors and the clinical status of CP-receiving patients according to the modified WHO 6-point ordinal scale
Impact of anti-SARS-CoV-2 antibody levels in donors on the viral clearance in CP-receiving patients | Days 0, 3, 6, 14, 21, and 28
  Correlation between anti-SARS-CoV-2 antibody levels in the donors and the viral clearance in CP-receiving patients. Additional test on day 3 will be performed to identify the early clearance of the virus.

CONTACTS AND LOCATIONS:
Overall Officials: David H Muljono, MD, PhD., Principal Investigator — Eijkman Institute for Molecular Biology; Irmansyah, MD, PhD, Principal Investigator — National Institute of Health Research and Development, Ministry of Health Republic of Indonesia; Sri Idaiani, MD, PhD, Study Director — National Institute of Health Research and Development, Ministry of Health Republic of Indonesia; Tetra Fajarwati, MD,PhD, Study Director — National Institute of Health Research and Development, Ministry of Health Republic of Indonesia
Locations (28):
- Indonesia (28):
  - Sanglah Central Hospital, Denpasar, Bali
  - Udayana University Hospital, Denpasar, Bali
  - Dr. Soeradji Tirtonegoro Hospital, Klaten, Central Java
  - Dr. Wongsonegoro Regency Hospital, Semarang, Central Java
  - Pasar Minggu Hospital, Jakarta, DKI
  - Dr. Haryoto Regency Hospital, Lumajang, East Java
  - Waluyo Jati Kraksaan Regency Hospital, Probolinggo, East Java
  - Sidoarjo Regency Hospital, Sidoarjo, East Java
  - Dr Ramelan Navy Hospital, Surabaya, East Java
  - Dr. Soetomo Hospital, Surabaya, East Java
  - Emergency Hospital for COVID-19 - Wisma Atlet Kemayoran, Jakarta Pusat, Jakarta Special Capital Region
  - Prof. Dr. R.D. Kandou Hospital, Manado, North Sulawesi
  - Dr. Tadjuddin Chalid Hospital, Makassar, Souh Sulawesi
  - Dr. Wahidin Sudirohusodo Central Hospital, Makassar, South Sulawesi
  - Hasanuddin University Hospital, Makassar, South Sulawesi
  - Dadi Hospital, Makassar, South Sulawesi
  - Dr. Mohammad Hoesin Central Hospital, Palembang, South Sumatra
  - Aceh Tamiang Hospital, Aceh Tamiang, Special Region of Aceh
  - Dr. Hasan Sadikin Central Hospital, Bandung, West Java
  - RSD Gunung Jati, Cirebon, West Java
  - dr. Cipto Mangunkusumo National Central General Hospital, Jakarta
  - YARSI Hospital, Jakarta
  - Dr. Suyoto Pusrehab Kemenhan Hospital, Jakarta
  - Persahabatan Central hospital, Jakarta
  - Fatmawati Central Hospital, Jakarta
  - Prof. Dr. Sulianti Saroso Infectious Disease Hospital, Jakarta
  - University Of Indonesia Hospital (RSUI), Jakarta
  - Gatot Soebroto Central Army Hospital, Jakarta Pusat

IPD SHARING:
Plan to Share IPD: Yes
The original datasets used for this study are not publicly available due to the existing regulation, and only can be shared upon the approval of the Sponsor on behalf of the Ministry of Health.
Supporting Information: Study Protocol
Time Frame: January 1 - December 31, 2021
Access Criteria: The study protocol and and raw data are only shared to the ClinicalTrials.gov and/or Journal Reviewers.

REFERENCES:
- [Background] Casadevall A, Pirofski LA. The convalescent sera option for containing COVID-19. J Clin Invest. 2020 Apr 1;130(4):1545-1548. doi: 10.1172/JCI138003. No abstract available. PMID 32167489
- [Background] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- [Background] Li L, Zhang W, Hu Y, Tong X, Zheng S, Yang J, Kong Y, Ren L, Wei Q, Mei H, Hu C, Tao C, Yang R, Wang J, Yu Y, Guo Y, Wu X, Xu Z, Zeng L, Xiong N, Chen L, Wang J, Man N, Liu Y, Xu H, Deng E, Zhang X, Li C, Wang C, Su S, Zhang L, Wang J, Wu Y, Liu Z. Effect of Convalescent Plasma Therapy on Time to Clinical Improvement in Patients With Severe and Life-threatening COVID-19: A Randomized Clinical Trial. JAMA. 2020 Aug 4;324(5):460-470. doi: 10.1001/jama.2020.10044. PMID 32492084
- [Background] Szako L, Farkas N, Kiss S, Vancsa S, Zadori N, Vorhendi N, Eross B, Hegyi P, Alizadeh H. Convalescent plasma therapy for COVID-19 patients: a protocol of a prospective meta-analysis of randomized controlled trials. Trials. 2021 Feb 1;22(1):112. doi: 10.1186/s13063-021-05066-2. PMID 33522939
- [Background] Focosi D, Anderson AO, Tang JW, Tuccori M. Convalescent Plasma Therapy for COVID-19: State of the Art. Clin Microbiol Rev. 2020 Aug 12;33(4):e00072-20. doi: 10.1128/CMR.00072-20. Print 2020 Sep 16. PMID 32792417
- [Background] Diago-Sempere E, Bueno JL, Sancho-Lopez A, Rubio EM, Torres F, de Molina RM, Fernandez-Cruz A, de Diego IS, Velasco-Iglesias A, Payares-Herrera C, Flecha IC, Avendano-Sola C, Palomino RD, Ramos-Martinez A, Ruiz-Antoran B. Evaluation of convalescent plasma versus standard of care for the treatment of COVID-19 in hospitalized patients: study protocol for a phase 2 randomized, open-label, controlled, multicenter trial. Trials. 2021 Jan 20;22(1):70. doi: 10.1186/s13063-020-05011-9. PMID 33472681
- [Background] WHO Working Group on the Clinical Characterisation and Management of COVID-19 infection. A minimal common outcome measure set for COVID-19 clinical research. Lancet Infect Dis. 2020 Aug;20(8):e192-e197. doi: 10.1016/S1473-3099(20)30483-7. Epub 2020 Jun 12. PMID 32539990
- [Background] Siddiqi HK, Mehra MR. COVID-19 illness in native and immunosuppressed states: A clinical-therapeutic staging proposal. J Heart Lung Transplant. 2020 May;39(5):405-407. doi: 10.1016/j.healun.2020.03.012. Epub 2020 Mar 20. No abstract available. PMID 32362390
- [Background] Borghesi A, Maroldi R. COVID-19 outbreak in Italy: experimental chest X-ray scoring system for quantifying and monitoring disease progression. Radiol Med. 2020 May;125(5):509-513. doi: 10.1007/s11547-020-01200-3. Epub 2020 May 1. PMID 32358689
- [Background] Ekmekci PE, Arda B. Interculturalism and Informed Consent: Respecting Cultural Differences without Breaching Human Rights. Cultura (Iasi). 2017;14(2):159-172. PMID 29645014
- [Background] Zulu JM, Sandoy IF, Moland KM, Musonda P, Munsaka E, Blystad A. The challenge of community engagement and informed consent in rural Zambia: an example from a pilot study. BMC Med Ethics. 2019 Jul 4;20(1):45. doi: 10.1186/s12910-019-0382-x. PMID 31272489
- [Background] Janiaud P, Axfors C, Schmitt AM, Gloy V, Ebrahimi F, Hepprich M, Smith ER, Haber NA, Khanna N, Moher D, Goodman SN, Ioannidis JPA, Hemkens LG. Association of Convalescent Plasma Treatment With Clinical Outcomes in Patients With COVID-19: A Systematic Review and Meta-analysis. JAMA. 2021 Mar 23;325(12):1185-1195. doi: 10.1001/jama.2021.2747. PMID 33635310
- [Background] Libster R, Perez Marc G, Wappner D, Coviello S, Bianchi A, Braem V, Esteban I, Caballero MT, Wood C, Berrueta M, Rondan A, Lescano G, Cruz P, Ritou Y, Fernandez Vina V, Alvarez Paggi D, Esperante S, Ferreti A, Ofman G, Ciganda A, Rodriguez R, Lantos J, Valentini R, Itcovici N, Hintze A, Oyarvide ML, Etchegaray C, Neira A, Name I, Alfonso J, Lopez Castelo R, Caruso G, Rapelius S, Alvez F, Etchenique F, Dimase F, Alvarez D, Aranda SS, Sanchez Yanotti C, De Luca J, Jares Baglivo S, Laudanno S, Nowogrodzki F, Larrea R, Silveyra M, Leberzstein G, Debonis A, Molinos J, Gonzalez M, Perez E, Kreplak N, Pastor Arguello S, Gibbons L, Althabe F, Bergel E, Polack FP; Fundacion INFANT-COVID-19 Group. Early High-Titer Plasma Therapy to Prevent Severe Covid-19 in Older Adults. N Engl J Med. 2021 Feb 18;384(7):610-618. doi: 10.1056/NEJMoa2033700. Epub 2021 Jan 6. PMID 33406353
- [Background] Marx R, Eggert G, Beldner W. [Thermal expansion and plasticizing temperatures of dental adhesives]. Dtsch Zahnarztl Z. 1988 Apr;43(4):465-8. No abstract available. German. PMID 3044747
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2009 Jan;32 Suppl 1(Suppl 1):S62-7. doi: 10.2337/dc09-S062. No abstract available. PMID 19118289
- [Background] Jones AE, Trzeciak S, Kline JA. The Sequential Organ Failure Assessment score for predicting outcome in patients with severe sepsis and evidence of hypoperfusion at the time of emergency department presentation. Crit Care Med. 2009 May;37(5):1649-54. doi: 10.1097/CCM.0b013e31819def97. PMID 19325482
- [Background] Wiesner R, Edwards E, Freeman R, Harper A, Kim R, Kamath P, Kremers W, Lake J, Howard T, Merion RM, Wolfe RA, Krom R; United Network for Organ Sharing Liver Disease Severity Score Committee. Model for end-stage liver disease (MELD) and allocation of donor livers. Gastroenterology. 2003 Jan;124(1):91-6. doi: 10.1053/gast.2003.50016. PMID 12512033
- [Background] Cholongitas E, Papatheodoridis GV, Vangeli M, Terreni N, Patch D, Burroughs AK. Systematic review: The model for end-stage liver disease--should it replace Child-Pugh's classification for assessing prognosis in cirrhosis? Aliment Pharmacol Ther. 2005 Dec;22(11-12):1079-89. doi: 10.1111/j.1365-2036.2005.02691.x. PMID 16305721
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Oct 15;62(16):e147-239. doi: 10.1016/j.jacc.2013.05.019. Epub 2013 Jun 5. No abstract available. PMID 23747642
- [Background] Ng JJ, Luo Y, Phua K, Choong AMTL. Acute kidney injury in hospitalized patients with coronavirus disease 2019 (COVID-19): A meta-analysis. J Infect. 2020 Oct;81(4):647-679. doi: 10.1016/j.jinf.2020.05.009. Epub 2020 May 8. No abstract available. PMID 32389782
- See also: Convalescent Plasma for COVID-19. A randomized clinical trial — https://www.medrxiv.org/content/10.1101/2020.07.01.20139857v1
- See also: Clinical management of COVID-19: Interim guidance — https://www.who.int/publications/i/item/clinical-management-of-covid-19/
- See also: NCI Common Terminology Criteria for Adverse Events (CTCAE) — https://evs.nci.nih.gov/ftp1/CTCAE/About.html